CLINICAL TRIAL: NCT01624805
Title: Phase II Study of Horse Anti-Thymocyte Globulin (hATG), Cyclosporine, Methylprednisolone, and GCSF (Filgrastim or Pegfilgrastim) in Patients With Aplastic Anemia (AA), or Low/Int-1 Risk Myelodysplastic Syndrome (MDS)
Brief Title: Methylprednisolone, Horse Anti-Thymocyte Globulin, Cyclosporine, Filgrastim, and/or Pegfilgrastim or Pegfilgrastim Biosimilar in Treating Patients With Aplastic Anemia or Low or Intermediate-Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0334; NCI-2012-01096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0334 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Aplastic Anemia; de Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome
MeSH Terms: conditions — Anemia, Aplastic; Myelodysplastic Syndromes | interventions — Antilymphocyte Serum; thymoglobulin; Cyclosporine; Cyclosporins; Filgrastim; Granulocyte Colony-Stimulating Factor; Methylprednisolone; exifone; Medrol Veriderm; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (methylprednisolone, hATG, cyclosporine, G-CSF) (Experimental): Patients receive methylprednisolone IV over 10 minutes on days 1-4 and IV or PO with taper over days 5-30. Patients also receive horse anti-thymocyte globulin IV over 8 hours daily on days 1-4, cyclosporine PO BID on days 1-180, and pegfilgrastim or pegfilgrastim biosimilar SC on day 5 and/or filgrastim SC beginning on day 5 and continuing until absolute neutrophil count recovers. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Cyclosporine; Biological: Filgrastim; Drug: Methylprednisolone; Biological: Pegfilgrastim

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Methylprednisolone — Given IV or PO
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; SD-01; SD-01 sustained duration G-CSF

SUMMARY:
This phase II trial studies methylprednisolone, horse anti-thymocyte globulin, cyclosporine, filgrastim, and/or pegfilgrastim or pegfilgrastim biosimilar in treating patients with aplastic anemia or low or intermediate-risk myelodysplastic syndrome. Horse anti-thymocyte globulin is made from horse blood and targets immune cells known as T-lymphocytes. Since T-lymphocytes are believed to be involved in causing low blood counts in aplastic anemia and in some cases of myelodysplastic syndromes, killing these cells may help treat the disease. Methylprednisolone and cyclosporine work to suppress immune cells called lymphocytes. This may help to improve low blood counts in aplastic anemia and myelodysplastic syndromes. Filgrastim and pegfilgrastim are designed to cause white blood cells to grow. This may help to fight infections and help improve the white blood cell count. Giving methylprednisolone and horse anti-thymocyte globulin together with cyclosporine, filgrastim, and/or pegfilgrastim may be an effective treatment for patients with aplastic anemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of the combination of hATG (horse anti-thymocyte globulin), methylprednisolone, cyclosporine, and GCSF (filgrastim) in achieving response (complete response [CR], partial response [PR], or hematologic improvement [HI]) in patients with aplastic anemia, or myelodysplastic syndromes (MDS).

SECONDARY OBJECTIVES:

I. To assess the safety, tolerability, and toxicities of the combination of hATG, methylprednisolone, cyclosporine, and GCSF in patients with aplastic anemia, or MDS. II. To assess time to response, response duration, and overall survival of patients with aplastic anemia, or MDS being treated with the combination of hATG, methylprednisolone, cyclosporine, and GCSF.

OUTLINE:

Patients receive methylprednisolone intravenously (IV) over 10 minutes on days 1-4 and IV or orally (PO) with taper over days 5-30. Patients also receive horse anti-thymocyte globulin IV over 8 hours daily on days 1-4, cyclosporine PO twice daily (BID) on days 1-180, and pegfilgrastim or pegfilgrastim biosimilar subcutaneously (SC) on day 5 and/or filgrastim SC beginning on day 5 and continuing until absolute neutrophil count recovers. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of MDS (Low, Int-1 by IPSS, or hypocellular) who are either previously treated or untreated are eligible for this trial.
2. Patients with the diagnosis of aplastic anemia who are either previously treated or untreated are eligible if they are not currently candidates for an allogeneic stem cell transplant.
3. Patients ages 18 years and older are eligible
4. Patients must have been off of cytotoxic, immunosuppressive (except steroids), or targeted therapy for at least 2 weeks prior to entering this study, and have recovered from the toxic effects of that therapy to grade 1 or less.
5. Adequate organ function as defined below:

   * liver function (bilirubin < 2mg/dL, AST <3 x ULN)
   * kidney function (creatinine < 2.5 x ULN ).
6. ECOG performance status of ≤ 2.
7. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
9. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.
10. Patients should have an indication for therapy for their disease such as transfusion dependence or morbidity associated with their cytopenia(s) such as bleeding, severe fatigue, or frequent/multiple infections (eg. neutropenia).

Exclusion Criteria:

1. Pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study agents, breastfeeding should be discontinued if the mother is treated on this study.
2. Known HIV infection.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patient with documented hypersensitivity to any of the component medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-06-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Achievement of response | Up to 6 years
  Measured by complete response (CR), partial response, or hematologic improvement.

SECONDARY OUTCOMES:
Time to response | The interval between treatment start and the date of response, assessed up to 6 years
  Estimated according to the Kaplan-Meier method.
Duration of CR | Time interval between the date of CR to the date of first evidence of disease recurrence or death, assessed up to 6 years
  Estimated according to the Kaplan-Meier method.
Overall survival | Time from treatment start until the death or last follow-up time, assessed up to 6 years
  Estimated according to the Kaplan-Meier method.
Incidence of adverse events | Up to 6 years
  Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Tabulated by grade and course of therapy. Numbers of required dose reductions will be included in the toxicity report.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org